CLINICAL TRIAL: NCT05893264
Title: Sonographic Predictors of Difficult Epidural Placement.
Acronym: PREC-EPI
Status: Withdrawn | Type: Observational
Why Stopped: Study has been withdrawn as after IRB approval PI changed his working institution making the conduction of the study unfeasible
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Alessandro De Cassai, Principal Investigator, University of Padova
Other Study IDs: PREC-EPI
Record Dates: First submitted 2023-05-29; First posted 2023-06-07 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Anesthesia; Safety Issues; Epidural; Anesthesia, Headache
Keywords: technique; epidural; predictors; placement
MeSH Terms: conditions — Headache | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Epidural placement: All patients undergoing epidural placement will be enrolled.
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Several data will be collected such as:
  Age, weight, height, gender, previous spine surgery, skoliosis (Y/N), palpable spinous process (Y/N), experience in years of anesthesiologist, spine level of epidural placement
  and the following sonographic parameters at the level of epidural placement: skin-spinous process distance (cm), skin-transversous process distance (cm), erector spinae plane distance (cm), superior to inferior spinous process distance (cm)

SUMMARY:
Epidural placement is a commonly used procedure for pain management during labor, delivery, and surgeries. However, epidural placement is often considered a technically challenging and complex procedure that requires a high level of skill and experience. In cases where the epidural is improperly placed or fails to produce effective analgesia, the discomfort and distress experienced by the patient may be heightened. Hence, the use of predictors, such as sonographic ones, may prove to be a valuable tool for healthcare professionals in the placement of epidurals, ultimately ensuring successful pain management for patients.

The present study aims to identify predictors of difficult epidural placement in patients undergoing surgery.

ELIGIBILITY:
Inclusion Criteria:

* Surgery with epidural placement
* Age > 18 years

Exclusion Criteria:

* patient refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients undergoing surgery with epidural analgesia or anesthesia
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-08-14 (Actual); Primary Completion 2023-08-14 (Actual); Study Completion 2023-08-14 (Actual)

PRIMARY OUTCOMES:
Incidence of difficult epidural placement | through study completion, an average of 2 year
  Described as the requirement to replace the needle by fully removing it from the skin.

SECONDARY OUTCOMES:
Total body weight (kg) as predictive parameter for difficult epidural placement | through study completion, an average of 2 year
  Total body weight (kg) as predictive parameter for difficult epidural placement
Age (years) as predictive parameter for difficult epidural placement | through study completion, an average of 2 year
  Age (years) as predictive parameter for difficult epidural placement
Height (cm) as predictive parameter for difficult epidural placement | through study completion, an average of 2 year
  Height (cm) as predictive parameter for difficult epidural placement
Palpable spinous process (well, not well, not palpable) as predictive parameter for difficult epidural placement | through study completion, an average of 2 year
  Palpable spinous process (well, not well, not palpable) as predictive parameter for difficult epidural placement
Previous spine surgery (yes, no) as predictive parameter for difficult epidural placement | through study completion, an average of 2 year
  Previous spine surgery (yes, no) as predictive parameter for difficult epidural placement
Anesthesiology experience (years) as predictive parameter for difficult epidural placement | through study completion, an average of 2 year
  Anesthesiology experience (years) as predictive parameter for difficult epidural placement
Sonographic skin to spinous process distance(cm) as predictive parameter for difficult epidural placement | through study completion, an average of 2 year
  Sonographic skin to spinous process distance (cm) as predictive parameter for difficult epidural placement
Sonographic spinous process to spinous process distance (cm)as predictive parameter for difficult epidural placement | through study completion, an average of 2 year
  Sonographic spinous process to spinous process distance (cm)as predictive parameter for difficult epidural placement
Sonographic skin to transverse process distance (cm) as predictive parameter for difficult epidural placement | through study completion, an average of 2 year
  Sonographic skin to transverse process distance (cm) as predictive parameter for difficult epidural placement
Sonographic erector spine muscle group size (cm) as predictive parameter for difficult epidural placement | through study completion, an average of 2 year
  Sonographic erector spine muscle group size (cm) as predictive parameter for difficult epidural placement

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Padova, Padua, Veneto, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Data could be shared after ethical committee clearence and on a reasonable request